CLINICAL TRIAL: NCT00866333
Title: A Phase 2 Multi-Center Study of Entinostat (SNDX-275) in Patients With Relapsed or Refractory Hodgkin's Lymphoma
Brief Title: A Phase 2 Multi-Center Study of Entinostat (SNDX-275) in Patient With Relapsed or Refractory Hodgkin's Lymphoma
Acronym: ENGAGE-501
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated prior to completion of accrual per corporate decision.
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-275-0501
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; Relapsed Hodgkin's Lymphoma; Refractory Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — entinostat

STUDY DESIGN:
Intervention Model Description: The Single Group Assignment is one of three regimens based on the protocol version at the time of enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entinostat (Experimental): Regimen determined by protocol version.
  Regimen 1: entinostat 10 mg (two 5 mg tablets) orally, once every two weeks (Days 1 and 15) in a 28-day cycle until disease progression or unacceptable toxicity.
  Regimen 2: entinostat 10 mg (two 5 mg tablets) orally on Day 1, increased to 15 mg (three 5 mg tablets) beginning on Day 15 of Cycle 1 for participants who had not experienced treatment-related adverse events with severity grade ≥2 (moderate), then continue 15 mg every two weeks (Days 1 and 15) in a 28-day cycle until disease progression or unacceptable toxicity.
  Regimen 3: entinostat 15 mg (three 5 mg tablets), orally, once weekly for 3 weeks followed by a 1-week break in a 4-week (28-day) cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Entinostat

INTERVENTIONS:
Drug: Entinostat — Entinostat tablets
  Other Names: SNDX-275

SUMMARY:
This study will evaluate the efficacy and safety of entinostat, SNDX-275, in patients with relapsed or refractory Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic confirmation of relapsed or refractory classical Hodgkin's lymphoma from the last biopsy available. Relapsed disease is defined as progressive disease following systematic therapy(ies) with curative intent. Refractory disease is defined as disease not responding to or having progressed within 3 months of the last dose of most recent systemic therapy.
2. Must have progressed after, or been ineligible for, stem cell transplantation.
3. Documented disease that is radiographically measurable (≥ 1.5 cm in the largest transverse dimension). If only 1 site of radiographically measurable lesion with the longest diameter < 2.5 cm, lesion must be positive by Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) or biopsy.
4. Last dose of cytotoxic chemotherapy must be > 21 days before the first dose of study drug.
5. European Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Age 18 years or older.
7. Total Bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) and Aspartate Transaminase (AST) and Alanine Transaminase (ALT) ≤ 2.5 x ULN, possible exceptions if documented Hodgkin Lymphoma (HL) liver involvement.
8. Serum Creatinine ≤ 1.5 x ULN.
9. Absolute neutrophil counts of ≥ 1,000/µL, and platelet counts ≥ 50,000/µL
10. Patients or their legal representative must be able to read, understand, and sign a written informed consent

Exclusion Criteria:

1. Patients with another active cancer (excluding basal cell carcinoma or CIN/cervical carcinoma in situ or melanoma in situ). Prior history of other cancer is allowed, excluding active disease within the prior 5 years.
2. Prior allogeneic stem cell transplantation requiring active immunosuppressive therapy within 3 months of registration or with evidence of active Graft Versus Host Disease (GVHD).
3. Pregnant or lactating women. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test prior to start of study drug.
4. WOCBP and men whose partners are WOCBP must use an acceptable method of contraception while enrolled on this study, and for a period of 3 months following the last dose of study drug.
5. Patients with uncontrolled intercurrent illness, active or uncontrolled infections, or a fever > 38.5⁰C that has not been evaluated for infection on the day of scheduled dosing.
6. Patients who have been treated with any investigational drug within 28 days prior to the first dose of study medication, or who are receiving concurrent treatment with other experimental drugs or anti-cancer therapy.
7. Prior treatment with Histone Deacetylase (HDAC) inhibitors (e.g. valproic acid, Zolinza (SAHA), romidepsin (Istodax),and experimental compounds such as MethylGene's MCGD0103 and Novartis' LBH589).
8. History of pericarditis or pericardial effusion that had required medical or surgical intervention in the last 6 months, or myocardial infarction or arterial thromboembolic events within 6 months, or experiencing severe or unstable angina, or New York Heart Association (NYHA) Class III or IV disease or a QTc interval >0.47 seconds.
9. Known human immunodeficiency virus (HIV) or a history of active Hepatitis B or C as evidenced by laboratory abnormalities in addition to positive serology.
10. Active central nervous system lymphoma and lymphoma with leptomeningeal involvement.
11. Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc) that, in the judgment of the investigator, may affect the patient's ability to sign the informed consent and comply with study procedures.
12. Any condition that will put the patient at undue risk or discomfort as a result of adherence to study procedures.
13. History of gastrointestinal disorders (medical disorder or extensive surgery) that could interfere with absorption of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-04-13; Primary Completion 2013-02-08 (Actual); Study Completion 2013-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - University of Colorado, Denver, Colorado
  - Johns Hopkins, Baltimore, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Batlevi CL, Kasamon Y, Bociek RG, Lee P, Gore L, Copeland A, Sorensen R, Ordentlich P, Cruickshank S, Kunkel L, Buglio D, Hernandez-Ilizaliturri F, Younes A. ENGAGE- 501: phase II study of entinostat (SNDX-275) in relapsed and refractory Hodgkin lymphoma. Haematologica. 2016 Aug;101(8):968-75. doi: 10.3324/haematol.2016.142406. Epub 2016 May 5. PMID 27151994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States from 13 April 2009 to 8 February 2013.
Pre-assignment Details: Participants with a diagnosis of Relapsed or Refractory Hodgkin's Lymphoma (HL) were enrolled into one of three entinostat dosing regimens based on the version of the protocol at their time of enrollment in the study.
Groups:
- Regimen 1: Entinostat 10 mg: Regimen 1: entinostat 10 mg (two 5 mg tablets) orally, once every two weeks (Days 1 and 15) in a 28-day cycle until disease progression or unacceptable toxicity.
- Regimen 2: Entinostat 10 mg/15 mg: Regimen 2: entinostat 10 mg (two 5 mg tablets) orally on Day 1, increased to 15 mg (three 5 mg tablets) beginning on Day 15 of Cycle 1 for participants who had not experienced treatment-related adverse events with severity grade ≥2 (moderate), then continue 15 mg every two weeks (Days 1 and 15) in a 28-day cycle until disease progression or unacceptable toxicity.
- Regimen 3: Entinostat 15 mg: Regimen 3: entinostat 15 mg (three 5 mg tablets), orally, once weekly for 3 weeks followed by a 1-week break in a 4-week (28-day) cycle until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Regimen 1: Entinostat 10 mg | Regimen 2: Entinostat 10 mg/15 mg | Regimen 3: Entinostat 15 mg
Started | 16 | 17 | 16
Completed | 11 | 10 | 4
Not Completed | 5 | 7 | 12
Not completed — Withdrawal of consent | 0 | 1 | 2
Not completed — Reason not Specified | 3 | 1 | 1
Not completed — Study Terminated by Sponsor | 2 | 5 | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1: Entinostat 10 mg | Regimen 2: Entinostat 10 mg/15 mg | Regimen 3: Entinostat 15 mg | Total
Number analyzed (Participants) | 16 | 17 | 16 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (10.33) | 37.4 (13.53) | 34.8 (10.31) | 35.0 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 10 | 24
  Male | 7 | 12 | 6 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1
  Black or African American | 2 | 0 | 0 | 2
  White | 10 | 17 | 15 | 42
  Other | 3 | 0 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Overall Response Based on the Participant's Best Response That is Documented Within the First 6 Cycles of Protocol Therapy
Description: Best Overall Response was defined as Complete Response (CR) or Partial Response (PR). Tumor response was assessed by the Investigators using the International Working Group revised response criteria for malignant lymphoma (Cheson, Pfistner et al. 2007). CR was defined as complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities definitely assignable to HL. PR was defined as: At least a 50% decrease in sum of the products of the greatest diameters (SPD) of the six largest dominant nodes or nodal masses, No increase in the size of other nodes, No new sites of disease.
Time Frame: Up to 6 months
Population: Per-Protocol (PP) population included all participants who met all of the following criteria: Completed at least 2 cycles of entinostat therapy and Underwent computed tomography (CT) or positron emission tomography (PET) scans at Screening and Day 1 of Cycle 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regimen 1: Entinostat 10 mg | Regimen 2: Entinostat 10 mg/15 mg | Regimen 3: Entinostat 15 mg
Number analyzed (Participants) | 12 | 17 | 12
percentage of participants | 8.3 [0.2 to 38.5] | 11.8 [1.5 to 36.4] | 16.7 [2.1 to 48.4]

2. Secondary Outcome: Percentage of Participants With Best Overall Response Based on the Participant's Best Response Documented Through the Entire Course of Protocol Therapy
Description: as for outcome 1
Time Frame: Regimen 1 and 2 median follow-up 36.6 months; Regimen 3 median follow-up 18.4 months
Population: PP population included all participants who met all of the following criteria: Completed at least 2 cycles of entinostat therapy and Underwent CT or PET scans at Screening and Day 1 of Cycle 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regimen 1: Entinostat 10 mg | Regimen 2: Entinostat 10 mg/15 mg | Regimen 3: Entinostat 15 mg
Number analyzed (Participants) | 12 | 17 | 12
percentage of participants | 8.3 [0.2 to 38.5] | 17.6 [3.8 to 43.4] | 16.7 [2.1 to 48.4]

3. Secondary Outcome: Duration of Objective Response for Participants Achieving CR or PR
Description: Duration of objective response was defined as the number of days from the start date of CR or PR (whichever status is recorded first), until the first date that recurrent or progressive disease was objectively documented.
Time Frame: Regimen 1 and 2 median follow-up 36.6 months; Regimen 3 median follow-up 18.4 months
Population: PP population included all participants who met all of the following criteria: Completed at least 2 cycles of entinostat therapy and Underwent CT or PET scans at Screening and Day 1 of Cycle 3. Analysis included all participants who achieved CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regimen 1: Entinostat 10 mg | Regimen 2: Entinostat 10 mg/15 mg | Regimen 3: Entinostat 15 mg
Number analyzed (Participants) | 1 | 3 | 2
months | NA [NA to NA] — Median, Lower and Upper Confidence Interval (CI) were not estimable because there were no participants with CR or PR who progressed. | 28.6 [20.2 to 28.6] | 8.3 [NA to NA] — Lower and Upper CI were not estimable because there was only 1 participant with CR or PR who progressed.

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) and Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A Treatment-Emergent Adverse Event (TEAE) is an AE that occurred after receive study drug. Any changes from baseline in vital signs, electrocardiogram results, and laboratory parameters assessed by the investigator to be clinically significant were reported as AEs. A SAE is defined as an AE that: is fatal, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity is a congenital anomaly/birth defect, is another significant medical hazard, such as new malignancy.
Time Frame: First dose to within 30 days of the last dose of study drug (Up to 34 months)
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1: Entinostat 10 mg | Regimen 2: Entinostat 10 mg/15 mg | Regimen 3: Entinostat 15 mg
Number analyzed (Participants) | 16 | 17 | 16
Participants
  Any TEAE | 16 | 17 | 16
  SAE | 2 | 7 | 3

ADVERSE EVENTS:
Time Frame: First dose of study drug to within 30 days of last dose (Up to 34 months)
Arm/Group | Regimen 1: Entinostat 10 mg | Regimen 2: Entinostat 10 mg/15 mg | Regimen 3: Entinostat 15 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 1/16
Serious Adverse Events (participants affected / at risk) | 2/16 | 7/17 | 3/16
Other Adverse Events (participants affected / at risk) | 16/16 | 17/17 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1: Entinostat 10 mg (N=16) | Regimen 2: Entinostat 10 mg/15 mg (N=17) | Regimen 3: Entinostat 15 mg (N=16)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0
Lung infection pseudomonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Subdural haemorrhage (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1: Entinostat 10 mg (N=16) | Regimen 2: Entinostat 10 mg/15 mg (N=17) | Regimen 3: Entinostat 15 mg (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 11 | 12
Anaemia (Blood and lymphatic system disorders) | 9 | 9 | 10
Neutropenia (Blood and lymphatic system disorders) | 9 | 6 | 9
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 12 | 7
Constipation (Gastrointestinal disorders) | 5 | 7 | 3
Vomiting (Gastrointestinal disorders) | 3 | 10 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 8 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Dysgeusia (Gastrointestinal disorders) | 0 | 1 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0
Oral candidiasis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0
Tooth abscess (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia klebsiella (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 7 | 7 | 5
Oedema peripheral (Hepatobiliary disorders) | 5 | 7 | 3
Pyrexia (General disorders) | 3 | 7 | 3
Chills (General disorders) | 2 | 3 | 3
Asthenia (General disorders) | 1 | 2 | 1
Pain (General disorders) | 1 | 2 | 0
Gait disturbance (General disorders) | 1 | 0 | 1
Catheter thrombosis (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Condition aggravated (General disorders) | 0 | 0 | 1
Crepitations (General disorders) | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Mucosal dryness (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Pitting oedema (General disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Contusion (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin candida (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 6 | 4
Dizziness (Nervous system disorders) | 0 | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Critical illness polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 2
Platelet count decreased (Investigations) | 1 | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1
Breath sounds abnormal (Nervous system disorders) | 1 | 0 | 1
Haemoglobin decreased (Nervous system disorders) | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 0
Weight increased (Investigations) | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 0
Blood creatinine (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Eosinophil percentage increased (Investigations) | 0 | 0 | 1
International normalised ratio decreased (Investigations) | 1 | 0 | 0
Monocyte count increased (Investigations) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 3 | 3
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Pericardial rub (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 2 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 0
Transfusion reaction (Immune system disorders) | 0 | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Ear infection (Ear and labyrinth disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the multi-center Study shall not be made before the first multi-site publication by Sponsor or Publications Committee. No Public Presentation by Institution or Investigator will be made until Study Documentation/Results from all sites are received and analyzed by Sponsor. Separate publication by Investigator will be delayed for a period of 18 months until the initial publication by Committee or Sponsor, or a determination is made not to make such publication.